CLINICAL TRIAL: NCT06683651
Title: A Multicenter, Randomized, Double-Masked, Placebo-Controlled Parallel Group Phase III Study to Evaluate the Efficacy and Safety of STN1013800 Ophthalmic Solution in Chinese Patients With Acquired Blepharoptosis
Brief Title: A Study in Chinese Patients With Acquired Blepharoptosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101380002CN
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Blepharoptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STN1013800 ophthalmic solution (Experimental): 0.1% STN1013800 ophthalmic solution administered once daily
  Interventions: Drug: STN1013800 ophthalmic solution
- STN1013800 ophthalmic solution Liquid Base, without STN1013800 (Placebo Comparator): STN1013800 ophthalmic solution Liquid Base, without STN1013800 administered once daily
  Interventions: Drug: STN1013800 ophthalmic solution Liquid Base, without STN1013800

INTERVENTIONS:
Drug: STN1013800 ophthalmic solution — Investigational Product: 0.1% STN1013800 ophthalmic solution
  Arms: STN1013800 ophthalmic solution
Drug: STN1013800 ophthalmic solution Liquid Base, without STN1013800 — Placebo control: STN1013800 ophthalmic solution Liquid Base, without STN1013800
  Arms: STN1013800 ophthalmic solution Liquid Base, without STN1013800

SUMMARY:
This is a Phase III Study to evaluate the efficacy and safety of STN1013800 Ophthalmic Solution in Chinese Patients with Acquired Blepharoptosis.

At present, there are no medicines for the treatment of acquired blepharoptosis in China.

Therefore, to evaluate the efficacy and safety of 0.1% STN1013800 ophthalmic solution, Vehicle (Placebo) are designed.

For the screening period, 3-7 days were set to confirm the subjects and judge their qualification. Dosage and administration were based on prior clinical trial results approved at 0.1% once daily for 42 days treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least one eye diagnosed with acquired blepharoptosis and presence of all the following criteria at screening:

  * Loss of reliable Leicester Peripheral Field Test (LPFT) of ≥ 8 points in the top 2 rows (LPFT Eligibility Score); subjects had to see at least 9 total points in the top 4 rows (LPFT Total Score).
  * This criterion had to be met in both the Visit 1 Hour 0 (V1H0) and Visit 1 Hour 6 (V1H6) LPFT assessments.
  * There had to be ≤4 points of variance between the V1H0 and the V1H6 LPFT Eligibility Score.
  * The Marginal Reflex Distance-1 (MRD-1), the distance from the pupil center to the margin of upper lid, ≤ 2 mm (no visible pupil center defaults to 0) in the same eye
  * Visual acuity is 0.25 decimals (i.e., Snellen 20/80) or better according to standard logarithmic visual acuity chart in the same eye
* Presence of all the following criteria at baseline:

  * Loss of reliable LPFT of ≥8 points in the top 2 rows (LPFT Eligibility Score) in the same eye; subjects had to see at least 9 total points in the top 4 rows (LPFT Total Score).
  * This criterion had to be met in the Visit 2 Hour 0 (V2H0) LPFT assessment
  * There had to be ≤4 points of variance between the V1H6 and the V2H0 LPFT Eligibility Score;
  * The MRD-1, the distance from the pupil center to the margin of upper lid, ≤ 2 mm (no visible pupil center defaults to 0) in the same eye
  * Visual acuity is 0.25 decimals (i.e., Snellen 20/80) or better according to standard logarithmic visual acuity chart in the same eye
* Female subjects are 1-year postmenopausal, surgically sterilized, or females of childbearing potential (females who had started their menstrual cycles) with a negative urine pregnancy test at screening. Females of childbearing potential had to use an acceptable form of contraception throughout the study.

Exclusion Criteria: In the study eye

* Dermatochalasis that extended less than 3 mm above the upper eyelid margin.
* Pseudoptosis (upper eyelid dermatochalasis that overhung the upper eyelid margin).
* In either eye: Congenital ptosis; Horner syndrome; Marcus Gunn jaw-winking syndrome; Myasthenia gravis.
* Mechanical ptosis, including ptosis due to orbital or lid tumour, cicatricial processes affecting the movements of the upper lid, and enophthalmos.
* Previous ptosis surgery (previous blepharoplasty [only] was allowed provided the surgery took place > 3 months prior to screening).
* Lid position affected by lid or conjunctival scarring; Visual field loss from any cause other than ptosis; History of herpes keratitis.
* History of closed/narrow angle glaucoma (unless patent peripheral iridotomy had been performed > 3 months prior to screening).
* Periocular neurotoxin (e.g., Botox®, Dysport®) injections within 3 months prior to screening and during the study.
* Topical application of bimatoprost (i.e., Latisse®) to the eyelashes within 7 days prior to screening and during the study.
* Use of topical ophthalmic medications including but not limited to anti-allergy [e.g., antihistamines like Emadine®, Patanol®], dry eye [e.g., Diquas®, Beifushu®; except artificial tears like Hyaluronate], antimicrobial drugs [e.g., antibiotics and antivirals like Cravit®,Tobrex®, Aciclovir], and anti-inflammatory drugs
* Current punctal plugs or placement of punctal plugs during the study.
* Current use of over-the-counter (OTC) vasoconstrictor/decongestant eye medication or any ophthalmic or non-ophthalmic α-adrenergic agonist including OTC products at any time during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean change from Baseline in the STN1013800 group versus the Vehicle (Placebo) group | Day 1 Hour 6 (Visit 2); Day 14 Hour 2 (Visit 3)
  Mean change from Baseline (Day 1, Hour 0) in the STN1013800 group versus the Vehicle (Placebo) group in number of points seen in the top 4 rows on the Leicester Peripheral Field Test (LPFT test) at 2 time points

SECONDARY OUTCOMES:
Mean change of margin reflex distance-1 (MRD-1) from Baseline in the STN1013800 group versus the Vehicle (Placebo) group | Day 1 Hour 6 (Visit 2); Day 14 Hour 2 (Visit 3)
  Mean change of MRD-1 from Baseline (Day 1, Hour 0) in the STN1013800 group versus the Vehicle (Placebo) group at 2 time points
Mean change of margin reflex distance-1 (MRD-1) from Baseline in the STN1013800 group versus the Vehicle (Placebo) group | Day 1 at Minute 5, Minute 15, Hour 2; Day 14 at Minute 5, Minute 15, Hour 6; Day 42 at Minute 5, Minute 15
  Mean change of MRD-1 from Baseline (Day1, Hour 0) in the STN1013800 group versus the Vehicle (Placebo) group at other timepoints

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Joint Shantou International Eye Center of Shantou University and the Chinese University of Hong Kong, Shantou, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The first affiliated hospital of Zhengzhou University, Zhengzhou, He'nan
  - The 2nd Affiliated Hospital of Harbin Medical University, Ha’erbin, Helongjiang
  - Wuhan Aier Eye Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The second norman bethune hospital of Jilin University, Changchun, Jilin
  - Dalian No.3 Peple's Hospital, Dali, Liaoning
  - The 4TH People's Hospital of Shenyang, Shenyang, Liaoning
  - Shandong Eye Hospital, Jinan, Shandong
  - Eye & Ent Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Eye Hospital, Taiyuan, Shanxi
  - Panzhihua Hospital of Integrated Chinese and Western Medicine, Panzhihua, Sichuan
  - Tianjin Eye Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital (SRRSH), affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Eye Hospital, Wenzhou Medical University / Zhejiang Eye Hospital, Wenzhou, Zhejiang